CLINICAL TRIAL: NCT07096466
Title: CELL REGENERATION EFFICACY
Brief Title: Skin Cell Regeneration Efficacy of Cosmetic Product
Acronym: Exfoliator
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Amazentis SA (Industry)
Collaborators: SGS proderm GmbH (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 25.0055-25
Record Dates: First submitted 2025-07-18; First posted 2025-07-31 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Healthy Skin

STUDY DESIGN:
Intervention Model Description: On each volar forearm two test areas (each sized 3 cm x 3 cm) will be defined. Test area 1 will denote the lower right, 2 the upper right forearm. Test areas 3 and 4 on left forearm will be allocated accordingly. Each forearm test area will undergo one of four treatments (stained or unstained with DHA; and treated or untreated with cosmetic product) so all four treatments are experienced by every participant. Overall, the four treatment conditions (one treatment per test area) will be:
  A) Untreated with cosmetic product, stained with DHA (negative control) B) Treated with cosmetic product, stained with DHA C) Untreated with cosmetic product, unstained (negative control) D) Treated with cosmetic product, unstained
  Treatments will be randomly and balanced assigned to the four volar forearm test areas.
  E) All participants will also apply two cosmetic products to the facial area.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Untreated, stained forearm (Experimental): On day 1, the volar forearm test area will undergo DHA staining (250μl of 10% DHA solution applied under occlusion with Finn Chambers for 8 hours). The cosmetic product will not be applied for two weeks to the volar forearm test area.
  Interventions: Other: DHA stain; Other: No cosmetic product application - forearm
- Treated, stained forearm (Experimental): On day 1, the volar forearm test area will undergo DHA staining (250μl of 10% DHA solution applied under occlusion with Finn Chambers for 8 hours). The cosmetic product will then be applied twice daily for two weeks to the volar forearm test area.
  Interventions: Other: DHA stain; Other: Cosmetic product application - forearm
- Untreated, unstained forearm (Experimental): On day 1, the volar forearm test area will not undergo DHA staining. The cosmetic product will not be applied for two weeks to the volar forearm test area.
  Interventions: Other: No DHA stain; Other: No cosmetic product application - forearm
- Treated, unstained forearm (Experimental): On day 1, the volar forearm test area will not undergo DHA staining. The cosmetic product will then be applied twice daily for two weeks to the volar forearm test area.
  Interventions: Other: No DHA stain; Other: Cosmetic product application - forearm
- Facial treatment (Experimental): For two weeks on the face (excluding eye area), a cleansing cosmetic product containing Mitopure will be applied twice daily, and the cosmetic test product (that is used on forearms) will be applied once daily.
  Interventions: Other: Cosmetic products application - face

INTERVENTIONS:
Other: DHA stain — On day 1, the volar forearm test area will undergo DHA staining (250μl of 10% DHA solution applied under occlusion with Finn Chambers for 8 hours)
  Arms: Treated, stained forearm; Untreated, stained forearm
Other: No DHA stain — On day 1, the volar forearm test area will not undergo DHA staining.
  Arms: Treated, unstained forearm; Untreated, unstained forearm
Other: Cosmetic product application - forearm — The cosmetic product will be applied twice daily for two weeks to the volar forearm test area.
  Arms: Treated, stained forearm; Treated, unstained forearm
Other: No cosmetic product application - forearm — The cosmetic product will not be applied for two weeks to the volar forearm test area.
  Arms: Untreated, stained forearm; Untreated, unstained forearm
Other: Cosmetic products application - face — For two weeks on the face (excluding eye area), a cleansing cosmetic product containing Mitopure will be applied twice daily, and the cosmetic test product (that is used on forearms) will be applied once daily.
  Arms: Facial treatment

SUMMARY:
The objective of the study is to investigate the effect of one cosmetic product (exfoliator) containing Mitopure on the skin cell regeneration as well as on the skin hydration and skin barrier function in comparison to an untreated control area on the volar forearms.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent to participate in the study
* Willingness to actively participate in the study and to come to the scheduled visits
* Female and/or male
* From 18 to 65 years of age
* Healthy skin in the test area
* Uniform skin color in the test area
* Fitzpatrick I-III
* Able to read and follow directions as outlined in the protocol

Exclusion Criteria:

* Female subjects: Pregnancy or lactation
* Drug addicts, alcoholics
* AIDS, HIV-positive or infectious hepatitis
* Conditions which exclude a participation or might influence the test reaction/evaluation
* Participation or being in the waiting period after participation in cosmetic and/or pharmaceutical studies pertaining to the test area
* Cancer not being diagnosed as cured and requiring chemotherapy, irradiation and/or hormonal treatment within the last 2 years
* Insulin-dependent diabetes mellitus (type 1 and 2)
* Documented allergies to cosmetic products and/or ingredients,
* Documented allergies to plaster systems or tape adhesives
* Active skin disease at the test area like acute dermatitis, that requires actual topical medication on the test area and/or systemic drug treatment according to a physician
* Wounds, moles, tattoos, scars, irritated skin, excessive hair growth, etc. at the test area that could influence the investigation
* All kinds of beard (except a moustache) during the whole study
* Any topical medication at the test area within the last 3 days prior to the start of the study and throughout the entire course of the study
* Topical medication with anti-inflammatories, antihistamines within 1 week prior to the start of the study
* Topical medication with Immuno-suppressive medication within 2 weeks prior to the start of the study
* Systemic (oral) medication with Antibiotic (except penicillin) or anti-inflammatory steroids within 4 weeks prior to the start of the study and throughout the entire course of the study
* Systemic (oral) medication with anti-inflammatory non-steroids within 2 weeks prior to the start of the study and throughout the entire course of the study
* Phototherapy within 4 weeks prior to the start of the study and throughout the entire course of the study
* Systemic (oral) medication with retinoids within 6 months prior to the start of the study and throughout the entire course of the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2025-06-23 (Actual); Primary Completion 2025-07-09 (Actual); Study Completion 2025-07-09 (Actual)

PRIMARY OUTCOMES:
Skin cell regeneration quantified by change in skin color measured by Chromameter (unit of measure: Individual Typological Angle; ITA°) | 14 days
  Skin cell regeneration is quantified by the change in skin colour. Skin colour is measured with the Chromameter instrument (skin colour unit of measure: Individual Typological Angle [ITA°]). Therefore, skin cell regeneration is measured by the change in ITA°, such that a larger positive change in ITA° represents improved skin cell regeneration. Skin cell regeneration will be calculated 4, 8, 11, and 14 days after baseline.

SECONDARY OUTCOMES:
Skin hydration | 14 days
  Change from baseline in skin hydration (assessed on skin capacitance by Corneometer) after 14 days.
Skin barrier function | 14 days
  Change from baseline in skin barrier function (assessed on Transepidermal water loss (TEWL) by Tewameter [g/(m²h)]) after 14 days.
Product traits | 14 days
  Subjective evaluation of product traits assessed via questionnaire after 14 days. Product traits will be assessed by the subjects with a list of closed questions with the following predefined identical options to tick:-2 = Fully disagree; -1 = Rather disagree; 1 = Rather agree; 2 = Fully agree

CONTACTS AND LOCATIONS:
Overall Officials: Dr Katrin Unbereit, Principal Investigator — SGS proderm GmbH
Locations (1):
- SGS proderm GmbH, Schenefeld, Germany

IPD SHARING:
Plan to Share IPD: No